CLINICAL TRIAL: NCT02050945
Title: The Effects of Physical Exercise Training in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Anders Rasmussen Rinnov, Administrator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H-2-2013-150
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: COPD; Exercise; Resistance Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Resistance Training; Exercise; Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with COPD (Experimental): Patients with COPD are to be trained 3 times a week for 8 weeks
  Interventions: Behavioral: Resistance training
- Control patients with COPD (Active Comparator): Control patients with COPD are to be trained 3 times a week for 8 weeks
  Interventions: Behavioral: Endurance training

INTERVENTIONS:
Behavioral: Resistance training
  Other Names: Strength training, skeletal muscle, exercise, muscle training
  Arms: Patients with COPD
Behavioral: Endurance training
  Arms: Control patients with COPD

SUMMARY:
The purpose of the present project is to investigate the physiological effects of two different types of exercise training in COPD patients. The patients will be examined before, during and after 8 weeks of training to evaluate the effect of different types of skeletal muscle stimulation on health related quality of life, 6 min walking distance, flow mediated dilation, and histological properties of skeletal muscle cells, regarding oxidative capacity, fiber type, purinergic receptor amounts and measures of systemic inflammation. The study will test the hypothesis that:

Resistance training is superior to endurance training in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC fixed ratio <0.70, FEV1: <60% of predicted and MRC > or equal to 3
* Arterial oxygen saturation at rest> 90%, BMI >18, LVEF> 45.
* Age: 40 - 80 years

The medical treatment will be continued unchanged during the study and additional prednisolone and /or antibiotic treatment will be prescribed in case of acute exacerbation.

Exclusion Criteria:

* Unstable ischemic heart disease, severe heart valve failure, pulmonary emboli, severe heart failure, severe infections, musculoskeletal disorders, malignant disease, contraindicated medicine as MAO inhibitors and anticoagulants.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle function | At baseline and after 8 weeks of traning
  Muscle biopsy

SECONDARY OUTCOMES:
Flow mediated dilation | Change from baseline at 8 weeks
  Endothelium function
Body composition | Change from baseline at 8 weeks
  DEXA scan
6 min walking test | Change from baseline at 8 weeks
Health Related Quality of Life - COPD assessment test (CAT) | Change from baseline at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Mortensen, DMSc, Study Chair — Centre of Inflammation and Metabolism, University of Copenhagen, Rigshospitalet
Locations (2):
- Denmark (2):
  - Centre of Physical Activity Resarch, Copenhagen, Capital Region
  - Centre of Physical Activity Research, Copenhagen, Capital Region